CLINICAL TRIAL: NCT03931629
Title: Study of the Efficiency and Workflow of Femtosecond Laser Assisted Cataract Surgery in a Spanish Public Hospital
Acronym: FLACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLACS
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-03

CONDITIONS: Cataract; Cataract Mature; Cataract, Nuclear
Keywords: FEMTOSECOND LASER; Femtosecond Laser-Assisted Cataract Surgery; CATARACT SURGERY; phacoemulsification; operation room workflow; public setting
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Study design. This study was composed of two phases and was carried out by three consultant surgeons. No resident or trainee was involved in the performance of the surgeries. In Phase I, one of the three surgeons operated the LensX®, another performed the FLACS surgery (FLACS I) in one operating room (OR1), while the third surgeon performed the conventional phacoemulsification procedure (MANUAL) in another operating room (OR2). On subsequent days, the surgeons rotated between LensX®, FLACS and MANUAL surgery (Figure 1). All the settings for the Infiniti® and the LensX® were the same for all surgeons (see below). The cataracts included in the FLACS I group were presumably straightforward, as they were part of the learning curve for the surgeons and were evaluated by consultant ophthalmologists (it must be considered that the maximum best-corrected visual acuity [BCVA] for being eligible for cataract surgery in the Andalusian public System is 0.4 logMAR).
Masking Description: NO MASKING
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CONVENTIONAL PHACO (Active Comparator): In Phase I, one of the three surgeons operated the LensX®, another performed the FLACS surgery (FLACS I) in one operating room (OR1), while the third surgeon performed the conventional phacoemulsification procedure (MANUAL) in another operating room (OR2). On subsequent days, the surgeons rotated between LensX®, FLACS and MANUAL surgery
  Interventions: Procedure: CONVENTIONAL PHACO
- FEMTOSECONDLASER (FLACS) (Active Comparator): In Phase I, one of the three surgeons operated the LensX®, another performed the FLACS surgery (FLACS I) in one operating room (OR1), while the third surgeon performed the conventional phacoemulsification procedure (MANUAL) in another operating room (OR2). On subsequent days, the surgeons rotated between LensX®, FLACS and MANUAL surgery
  Interventions: Procedure: CONVENTIONAL PHACO

INTERVENTIONS:
Procedure: CONVENTIONAL PHACO — Cataract surgery by means of Femtosecond Laser-Assisted Cataract Surgery,
  Other Names: FEMTOSECONDLASER (FLACS)

SUMMARY:
Purpose: To assess the time-efficiency of a designated operation room (OR) workflow in the introduction of Femtosecond laser-assisted cataract surgery (FLACS, LenSx, Alcon®). The study was carried out in a public hospital with high volume of procedures.

Setting: Ophthalmology department of a tertiary referral Spanish public hospital.

Design: Prospective, controlled, surgical intervention study. Methods: A total of 167 eyes were enrolled, including 62 eyes undergoing conventional phacoemulsification surgery. In phase I, patients were assigned either to FLACS-I (n=63) or conventional phacoemulsification surgery (n=62). One surgeon operated the Femto-second laser, another finished the procedure, whereas another performed a conventional phacoemulsification. In the second phase (FLACS-II), all the surgeries were FLACS (n=42). A surgeon performed the FLACS procedure and two different surgeons completed the surgeries in separated ORs. Surgical and roll-over times of all the patients were recorded.

DETAILED DESCRIPTION:
MATERIALS AND METHODS Patient recruitment. This single-center, prospective, consecutive, interventional, and non-randomized study was conducted at the Department of Ophthalmology of the Regional University Hospital of Málaga (Spain) from February to June 2016. Patients were recruited in this clinical setting during routine activity. Inclusion criteria for the study were signed informed consent, patients of more than 18 years old, presence of visually significant cataract (best corrected visual acuity worse than 0.4 logMAR), and possibility of performing cataract surgery under local anaesthesia (topical, sub-tenon or retrobulbar). Exclusion criteria were patients who refused to give their consent, traumatic, congenital, luxated, subluxated cataracts, or with manifest zonular weakness, vitrectomized patients, small pupils (mydriasis less than 6 mm), narrow palpebral fissure, advanced optic nerve glaucomatous excavation, irregular astigmatism, significant corneal opacities, severe ocular surface disease, keratoconus, stromal scarring or edema and patients requiring general anaesthesia for the intervention. Patients who complied with the inclusion and exclusion criteria mentioned above signed a specific informed consent for the study and were non-randomly assigned to the FLACS (femtosecond laser-assisted cataract surgery) or MANUAL (manual or conventional phacoemulsification surgery) group. We checked that both groups were comparable in terms of age and gender. The three surgeons involved in the study were highly experienced consultants in performing conventional cataract surgery (from 15 to 20 years of experience, performing from 500 to 800 phacoemulsifications yearly) and refractive surgery (10 to 15 years of experience, performing from 200 to 500 refractive procedures). This study has been carried out following the Declaration of Helsinki and Good Clinical Practices guidelines. Personal data was processed according to guidelines established by the Spanish Law of Data Protection (LOPD).

Study design. This study was composed of two phases and was carried out by three consultant surgeons. No resident or trainee was involved in the performance of the surgeries. In Phase I, one of the three surgeons operated the LensX®, another performed the FLACS surgery (FLACS I) in one operating room (OR1), while the third surgeon performed the conventional phacoemulsification procedure (MANUAL) in another operating room (OR2). On subsequent days, the surgeons rotated between LensX®, FLACS and MANUAL surgery (Figure 1). All the settings for the Infiniti® and the LensX® were the same for all surgeons (see below). The cataracts included in the FLACS I group were presumably straightforward, as they were part of the learning curve for the surgeons and were evaluated by consultant ophthalmologists (it must be considered that the maximum best-corrected visual acuity [BCVA] for being eligible for cataract surgery in the Andalusian public System is 0.4 logMAR). Patients with easily accessible sockets and good patient collaboration were included. Eligible cataracts ranged from nuclear opacities from NC1 to NC4, cortical opacities from C1 to C4 and posterior subcapsular from P1 to P4, according to the Lens Opacities Classifications System (LOCSIII); with good pupil dilation (minimum 8 mm, that was measured in the slit lamp as described by Ho et al29) after the standard dilation protocol, i.e., instillation of tropicamide 1% and fenylephrine 10% eye-drops in the conjunctival sac, three times, each time separated by 10 minutes. Fuchs endothelial dystrophy and white cataracts were excluded. To ensure the comparability among groups, cataracts included in the MANUAL group were selected with similar characteristics. In phase II, one of the three surgeons operated the LensX®, while the other two surgeons completed the procedures in two different ORs (FLACS II)(Figure 2). Surgeons rotated in subsequent days. The FLACS II group included patients with harder cataracts (nuclear opacities from NC4 to NC6, cortical opacities from C3 to C5 and posterior subcapsular from P3 to P5, according to the LOCSIII), smaller orbits, suboptimal mydriasis (from 6 to 8 mm, measured in the slit lamp as mentioned before), Fuchs endothelial dystrophy and white cataracts. (Images 1-3). Therefore, this group included the whole range of cataract surgeries that are commonly performed at a public hospital.

Procedures. Prior to surgery, the routine dilation protocol (instillation of tropicamide 1% and fenylephrine 10% eye-drops in the conjunctival sac, three times, each time separated by 10 minutes), preoperative disinfection (cleaning of eyelid and periorbital region with 10% povidone iodine and instillation of povidone iodine 5% in in the conjunctival sac) and placement of sterile dressing were performed as usual. Conventional phacoemulsification was performed using the divide-and-conquer technique through a 2.2-mm clear corneal incision and the platform Infiniti® (Alcon®, Fort Worth, Texas, USA). FLACS was performed using the LenSx® platform (Alcon® Fort Worth, Texas, USA). The femtosecond laser was placed in a room adjacent to the OR, complying with current sterility standards mentioned above. Patients were transported from the laser room to the OR in an ophthalmological surgical chair. After completing the laser-assisted procedures (capsulorrhexis, nucleus fragmentation, main and accessory incisions), the patient entered to the OR where the phacoemulsification and aspiration of the nucleus and cortical masses, implantation of the IOL (AcrySof® IQ Monofocal IOL, Alcon, Fort Worth, Texas, USA), and hydration of surgical borders were performed. The ophthalmic viscosurgical device used in all cases was DuoVisc® Alcon, Fort Worth, Texas, USA). Prophylactic 0.1 mL of cefuroxime (1 mg/0.1 mL) was injected in the anterior chamber at the end of the surgery. The postoperative follow-up was performed according to usual protocols.

Settings. All the settings for the Infiniti® and the LensX® were the same for all surgeons. The Infiniti® settings were the following: for the pre-phaco, 80 cmH20 of irrigation, 150 mmHg of vacuum and 25 mL/min of flow aspiration; for sculpt, 80 cmH20 of irrigation, 70% of phaco energy and 95% of torsional amplitude, 50 mmHg of vacuum and 25 mL/min of flow aspiration; for segment removal: 110 cmH20 of irrigation, 90 of torsional amplitude, 400 mmHg of vacuum and 25 mL/min of flow aspiration; for the epinucleus removal: 110 cmH20 of irrigation, 230 mmHg of vacuum and 25 mL/min of flow aspiration; for the irrigation/aspiration: 65 cmH20 of irrigation, 450 mmHg of vacuum and 25 mL/min of flow aspiration; for the visco 65 cmH20 of irrigation, 500 mmHg of vacuum and 30 mL/min of flow aspiration. Continous Ozil was used throughout the phacoemulsification. The settings for LensX® were the following. For the capsulotomy: diameter 5mm, energy 5 µJ, spot separation 4 µm, layer separation 3 µm, delta up (lens anterior offset) 300 µm, delta down (lens posterior offset) 300 µm. A three-plane incision was used for primary incision at 135 degrees (posterior depth 40, 80 and 130%, respectively). Secondary incision was performed at 45 degrees. For both incisions, energy used was 4 µJ and spot and layer separation was 4 µm. The laser pattern for fragmentation was a hybrid combination between chop (two cuts) and cylinder.

Measurements. The surgical and roll-over times for both conventional phacoemulsification and FLACS were recorded in a spreadsheet including: start time of patient preparation, start time of anesthesia, surgery start time, surgery end time, time needed to transfer the patient to resting area, and time of discharge. Specifically, for patients undergoing FLACS, the sum of the preparation time and the femtosecond laser time was calculated as well as the time between the performance of femtosecond laser procedures and the beginning of phacoemulsification surgery, and the time ranging from the moment when the patient entered to the femtosecond laser room to the moment where the patient left after the end of the surgery. Likewise, the following parameters were calculated in all groups: time from the insertion of blepharostat to its removal after ending the surgical procedure, time from the moment the patient entered the OR to the moment the patient left the OR after finishing the surgery, and time from the admission of the patient to the surgical area to the discharge once the intervention was finished. Likewise, mean phacoemulsification energy used in each procedure was also recorded (CDE: cumulative dissipated energy). Finally, intraoperative complications were also recorded, including loss of suction, loss of fixation/follow-up and incomplete capsulorrhexis for the femtosecond laser-assisted stage, and incomplete rexis, capsular rupture, IOL dislocation and incisions without coaptation for the phacoemulsification stage.

Statistical analysis. A descriptive analysis of the variables studied including mean, standard deviation, maximum and minimum. To analyse the differences between FLACS and MANUAL groups in terms of the continuous quantitative variables, the unpaired Student t test was applied whenever the normality condition was satisfied (verified with the Shapiro-Wilk test). Otherwise, the corresponding non-parametric test was used (Mann-Whitney test). Comparisons of categorical variables were performed using the Chi-square test. A homogeneity analysis was performed between groups in terms of age and gender to ensure the comparability of groups. All these statistical analyses were performed using R software version 3.2.1 (R Foundation for Statistical Computing, Vienna, Austria; available at http://www.R-project.org or R Development core Team, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signing.
* Over 18 years old.
* No medical contraindication for cataract surgery.
* Maximum best-corrected visual acuity [BCVA] 0.4 logMAR.
* Patients with easily accessible sockets.
* Minimal pupil mydriasis of 6 mm.
* Anticipated good patient collaboration.

Exclusion Criteria:

* No informed consent signing.
* Patients under 18 years old.
* Medical contraindication for cataract surgery.
* Maximum best-corrected visual acuity [BCVA] over 0.4 logMAR.
* Patients with badly accessible sockets.
* Maximal mydriasis inferior to 6 mm.
* Poor patient collaboration were included.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
WORKFLOW IN THE OPERATION ROOM (minutes) | Operation day
  Surgical and roll-over times (measured in minutes) for both conventional phacoemulsification and FLACS were assessed: start time of patient preparation, anesthesia and surgery, surgery end time, time needed to transfer the patient to resting area, and time of discharge; time from the insertion of blepharostat to its removal after ending the surgical procedure, time from the moment the patient entered the OR to the moment the patient left the OR after finishing the surgery, and time from the admission of the patient to the surgical area to the discharge once the intervention was finished.

SECONDARY OUTCOMES:
CUMULATIVE DISSIPATED ENERGY (MEASUREN IN %, PROVIDED BY THE PHACOEMULSIFICATION DEVICE) | Operation day
  Likewise, mean phacoemulsification energy values (measured in %, as provided bu the phacoemulsification device) used in each procedure was also recorded (CDE: cumulative dissipated energy).
INTRAOPERATIVE COMPLICATIONS | Operation day
  Intraoperative complications were also recorded, including loss of suction, loss of fixation/follow-up and incomplete capsulorrhexis for the femtosecond laser-assisted stage, and incomplete rexis, capsular rupture, IOL dislocation and incisions without coaptation for the phacoemulsification stage.

REFERENCES:
- [Derived] Villavilla-Castillo J, Perez-Casaseca C, Espejo-de-Los-Riscos E, Fernandez-Baca-Vaca G, Fernandez-Baca-Casares I, Pinero-Llorens DP, Rocha-de-Lossada C, Rodriguez-Calvo-de-Mora M. Study of the efficiency and workflow of femtosecond laser-assisted cataract surgery in a Spanish public hospital. J Fr Ophtalmol. 2021 Oct;44(8):1190-1201. doi: 10.1016/j.jfo.2021.01.030. Epub 2021 Jul 16. PMID 34275664